CLINICAL TRIAL: NCT00711984
Title: Comparison of Stenting Versus Best Medical Therapy for Treatment of Ostial Renal Artery Stenosis: a Randomized Controlled Trial in Patients With Advanced Atherosclerosis.
Brief Title: Comparison of Stenting Versus Best Medical Therapy for Treatment of Ostial Renal Artery Stenosis: a Trial in Patients With Advanced Atherosclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Erich Minar, Medical University Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0-2003
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Renal Artery Stenosis
Keywords: renal artery stenosis; stent; comparison of treatments; progression; atherosclerosis; peripheral artery disease; major cardiovascular events
MeSH Terms: conditions — Renal Artery Obstruction; Disease Progression; Atherosclerosis; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Renal artery stenting and Best medical treatment
  Interventions: Device: Herkulink renal artery Stent; Other: best medical therapy
- 2 (Active Comparator): Best medical treatment alone
  Interventions: Other: best medical therapy

INTERVENTIONS:
Device: Herkulink renal artery Stent — renal artery stent
  Other Names: Herkulink (renal stent) Guidant/Abbott Vascular
  Arms: 1
Other: best medical therapy — All patients will receive best medical therapy according to current guidelines consisting in antihypertensive, antiplatelet, antidiabetic and lipid-lowering medication and in recommendation of lifestyle modification

SUMMARY:
Renal artery stenosis (RAS) usually refers to a disease of the large extra-renal arterial vessels and most frequently is caused by atherosclerotic obstructions. The prevalence of atherosclerotic RAS increases with age, male gender, traditional cardiovascular risk factors (hypertension, diabetes, smoking, hyperlipidemia) and atherosclerotic comorbidities like coronary artery or peripheral artery disease (PAD). A prevalence up to 40% has been reported in patients with PAD. Undoubtedly, atherosclerotic RAS is a progressive disease, as more than half of the patients exhibit an increasing degree of stenosis within five years after diagnosis, and one out of five patients with a critical stenosis (>60%) suffers renal atrophy and renal failure during this period. RAS may be treated conservatively by so called best medical treatment, surgically, or by endovascular interventions using balloon angioplasty and stenting.

The purpose of the investigators study is to determine the incidence and the predictors of RAS in patients with PAD, and to compare the effect of renal artery stenting versus best medical treatment in patients with hypertension and ostial renal artery stenosis in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* PAD and unilateral ostial >60% RAS and hypertension

Exclusion Criteria:

* Conditions which imply RAS stenting (bilateral significant renal disease, single functioning kidney, or patients whose conditions cannot be managed medically or by intervention)
* Allergy to contrast agents or medication administered for best medical treatment (in particular ASA and statins)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-02

PRIMARY OUTCOMES:
change in mean blood pressure and renal function occurrence of major cardiovascular events | 3, 6, 9, 12 months, annually

SECONDARY OUTCOMES:
progression of the degree of RAS in the conservative group and restenosis rate in the stent group | 6, 12 months, annually

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria